CLINICAL TRIAL: NCT04505800
Title: Chrononutrition of Using L-tryptophan Supplementation to Alleviate the Impacts of Night Shift Rotation on Circadian Hormones and Health Outcomes
Brief Title: Tryptophan Supplementation to Improve Night Shift Workers' Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Hsin-Jen Chen, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: YM106114F
Record Dates: First submitted 2020-06-23; First posted 2020-08-10 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Sleep; Mood; Burnout; Melatonin Deficiency; Cortisol Deficiency
Keywords: tryptophan; shift work; randomized trial; melatonin; cortisol
MeSH Terms: conditions — Burnout, Psychological | interventions — Maltose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tryptophan supplement (Experimental): * Pure L-tryptophan in capsules (500mg/capsule)
  * 3g tryptophan per day (2 capsules, t.i.d.), at 8AM, 4PM, and 0AM (± 1 hour)
  Interventions: Dietary Supplement: Tryptophan supplement
- Maltose (Placebo Comparator): * Placebo is maltose powder capsule (500mg/capsule)
  * 3g maltose powder per day (2 capsules, t.i.d.), at 8AM, 4PM, and 0AM (± 1 hour)
  Interventions: Dietary Supplement: Maltose

INTERVENTIONS:
Dietary Supplement: Tryptophan supplement — * Pure L-tryptophan in capsules (500mg/capsule)
  * 3g tryptophan per day (2 capsules, t.i.d.), at 8AM, 4PM, and 0AM (± 1 hour)
  Arms: Tryptophan supplement
Dietary Supplement: Maltose — Maltose
  Arms: Maltose

SUMMARY:
This randomized cross-over double-blinded trial aims to investigate the health effect of oral l-tryptophan supplementation on workers who rotate night shift work, and to examine the influences of different frequencies and timings of supplementation on the health effects.

DETAILED DESCRIPTION:
This study aims to investigate the health effect of oral l-tryptophan supplementation on workers who rotate night shift work, and to examine the influences of different frequencies and timings of supplementation on the health effects. Night shift work affects melatonin and cortisol variation, insomnia, mood issues, and metabolic syndrome. Short-term tryptophan supplementation was shown to improve melatonin, sleep quality, and cortisol response to acute stress. Little is known whether a longer term of longer-term tryptophan supplementation would alleviate the health impacts of night shift work. Nevertheless, melatonin and cortisol have their normal circadian patterns. Nothing is known about what temporal structure of tryptophan supplement would maximize its health effects on night shift workers melatonin and cortisol levels. We will conduct a double-blind cross-over randomized controlled trial to examine the benefits of oral tryptophan administration (3g/day, t.i.d.) on night shift workers' health outcomes: melatonin and cortisol levels, sleep quality, moods and work performance. We expect to reveal the health effect of tryptophan supplementation in night shift workers by using sophisticated study design.

ELIGIBILITY:
Inclusion criteria:

* Age: adults >=20 y/o
* Adults who had night shift schedule >1 month before enrollment, and will have similar night shift schedule in the following 2 months. (Eligible night shift schedule: >1 day of evening or night shift in a week)
* People who will not have plans to travel to another time zone in the following 2-3 months
* People who will plan to stay in the same job position for the following 3 months
* People who have no experience in taking tryptophan or melatonin supplement in the past month
* Body weight >= 50kg and <=80kg
* Non-pregnant, non-breastfeeding, not taking contraceptives
* Not under treatment of steroids, not taking sleeping pills

Exclusion criteria:

* diagnosis of renal or liver diseases
* diagnosis of Cushing's Disease, Addison's disease
* psychiatric diagnosis, such as depression and anxiety disorders
* neurological diseases such as dementia, epilepsy, Parkinson's disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Melatonin level in the morning | 3 weeks
  Morning (8AM) saliva melatonin level change in the phase
Melatonin level in the afternoon | 3 weeks
  Afternoon (4PM) saliva melatonin level change in the phase
Melatonin level at midnight | 3 weeks
  Midnight (0AM) saliva melatonin level change in the phase
Cortisol level in the morning | 3 weeks
  Morning (8AM) saliva cortisol level change in the phase
Cortisol level in the afternoon | 3 weeks
  Afternoon (4PM) saliva cortisol level change in the phase
Cortisol level at midnight | 3 weeks
  Midnight (0AM) saliva cortisol level change in the phase

SECONDARY OUTCOMES:
Sleep quality | 3 weeks
  Pittsburg Sleep Quality Score (range: 0-21) at the end of the phase. The higher score indicates worse sleep quality
Mood states, depression | 3 weeks
  Depression, Anxiety, Stress Scales. Depression score (range 0-42) changes in the phase. The higher score, the more depressed.
Mood states, anxiety | 3 weeks
  Depression, Anxiety, Stress Scales. Anxiety score (range 0-42) changes in the phase. The higher score, the more anxious.
Mood states, stress | 3 weeks
  Depression, Anxiety, Stress Scales. Stress score (range 0-42) changes in the phase. The higher score, the more stressful.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The participants did not provide agreement to the researchers.